CLINICAL TRIAL: NCT06309160
Title: COMPASS Across Settings (CAST) for Integrating School, Home, and Community Services and Improving Transition Outcomes for Students With ASD
Brief Title: COMPASS Across Settings (CAST) for Improving Transition Outcomes for Students With ASD
Acronym: CAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Collaborators: University of Toledo (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A230008
Record Dates: First submitted 2024-01-22; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Autism; Autism Spectrum Disorder; Autistic Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Pre-post; randomized control
Who Masked: Outcomes Assessor
Masking Description: Independent observer evaluating goal attainment outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus Groups to Inform CAST (No Intervention): For the year 1 development activities, the research team will conduct focus groups with administrators, special education teachers, parents, students, and pre-employment transition specialists about how to integrate plans and services across settings.
- Pre-Post study of CAST (Experimental): The research team will then conduct a field test of CAST in year 2, making further revisions.
  Interventions: Behavioral: COMPASS Across Settings (CAST)
- Randomized Controlled Study of CAST (Active Comparator): In year 3, they will use a mixed methods design using a small RCT and network analysis, oversampling African American students and students from rural areas, to evaluate CAST for improved postsecondary outcomes in employment, training, and education.
  Interventions: Behavioral: COMPASS Across Settings (CAST)

INTERVENTIONS:
Behavioral: COMPASS Across Settings (CAST) — CAST will begin with an initial joint session with the student, caregiver, special education teacher, and pre-employment transition specialist that allows for discussion on the student's postsecondary goals, preferences, frustrations, challenges, and strengths related to social skills, adaptive/self-management, communication, problem behaviors, learning skills, and sensory sensitivities and preferences. This discussion will pinpoint critical social, communication, and work behavior/learning goals related to postsecondary goals and inform the intervention plans that are generated for each goal. Following this initial consultation, there will be four additional 1-hour sessions that incorporate evidence-based coaching, provided by the investigators, including performance feedback monitoring and instructional support. Each session is standardized and allows for assessment of student progress and intervention modification/self-reflection on the implementation of the intervention plans.
  Arms: Pre-Post study of CAST; Randomized Controlled Study of CAST

SUMMARY:
Purpose: The purpose of this project is to develop and test the COMPASS [Collaborative Model for Competence and Success] Across Settings (CAST) intervention to enhance the goal setting and attainment skills of autistic youth. Despite federal education law mandating transition services as part of the Individualized Education Program (IEP) for ensuring good outcomes for students with disabilities, current educational practices have been unable to demonstrate that autistic students experience positive postsecondary outcomes. There are existing, evidence-based interventions aimed at supporting positive outcomes for these students. However, these interventions have not systematically provided coaching support to the caregivers, students, and employment specialists. To address these issues, CAST will integrate three evidence-based interventions for supporting student transitions while providing this critical coaching support. By doing so, CAST aims to align the priorities and goals of interventions across home, school, and community settings to better support positive postsecondary outcomes for autistic students.

DETAILED DESCRIPTION:
Project Activities: The research team will use an iterative approach for integrating the three interventions into CAST, obtaining feedback from focus groups and stakeholder members along the way, and running a field trial after development. The research team will then conduct a randomized controlled trial (RCT) of CAST to examine postsecondary outcomes at both 3 months and 1 year after high school. Social network analysis will be used to understand the integration of services and a cost analysis will be conducted.

Products: This project will result in a fully developed intervention, CAST, for improving IEP and postsecondary outcomes of autistic students. The project will also result in peer-reviewed publications, information on the costs of CAST implementation, an updated intervention manual with fidelity checklists, and other dissemination products aimed at stakeholders.

STRUCTURED ABSTRACT

Setting: This project will take place in public high schools in Indiana.

Sample: Approximately 38 administrators, special education teachers, caregivers, pre-employment transition specialists, and autistic youth will participate in focus groups and interviews in the first year. The field test in year 2 will include five autistic youth and their parents, five classroom special education teachers, and five employment transition specialists. Approximately 140 participants (40 autistic youth and young adults, 40 caregivers, 40 special education teachers, and 20 pre-employment specialists who serve autistic youth) will participate in the pilot RCT in year 3.

Intervention: CAST will integrate three evidence-based interventions- COMPASS, C-HOPE, and COMPASS-T. COMPASS is the original intervention designed for preschool and elementary age students. COMPASS-T is the adaptation of COMPASS for transition-aged youth. Lastly, C-HOPE is based on COMPASS and is a parent-mediated intervention designed to decrease child problem behavior, increase parent competency, and decrease parent stress. CAST will begin with an initial joint session with the student, caregiver, special education teacher, and pre-employment transition specialist that allows for discussion on the student's postsecondary goals, preferences, frustrations, challenges, and strengths related to social skills, adaptive/self-management, communication, problem behaviors, learning skills, and sensory sensitivities and preferences. This discussion will pinpoint critical social, communication, and work behavior/learning goals related to postsecondary goals and inform the intervention plans that are generated for each goal. Following this initial consultation, there will be four additional 1-hour sessions that incorporate evidence-based coaching, provided by the investigators, including performance feedback monitoring and instructional support. Each session is standardized and allows for assessment of student progress and intervention modification/self-reflection on the implementation of the intervention plans.

Research Design and Methods: For the year 1 development activities, the research team will conduct focus groups with administrators, special education teachers, parents, students, and pre-employment transition specialists about how to integrate plans and services across settings. The research team will then conduct a field test of CAST in year 2, making further revisions. In year 3, they will use a mixed methods design using a small RCT and network analysis, oversampling African American students and students from rural areas, to evaluate CAST for improved postsecondary outcomes in employment, training, and education. The secondary aims of the project are to obtain (a) information on how well CAST improves integration and alignment of services across settings and thus student IEP and postsecondary outcomes; (b) information on feasibility, usability, and fidelity; and (c) estimates of costs.

Control Condition: Students in the control condition will receive services as usual.

Key Measures: The primary outcome data will be student goal attainment (GAS) of IEP goals and postsecondary goals. IEP goal attainment is assessed using psychometric equivalence goal attainment scaling (PET-GAS). Postsecondary outcomes will be assessed by parent report of attainment in goals (such as enrolling in a training or college program and living independently). Additional measures completed by all CAST participants (caregivers, students, special education teachers, and pre-employment specialists) include assessment of transition plan quality, organizational connectedness, and fidelity assessments.

Data Analytic Strategy: Focus groups and interviews will be recorded, transcribed, checked for accuracy, and analyzed using a consensual coding technique that will be used to provide a multi-dimensional picture for refining CAST. For the field test, the research team will use a dependent sample t-test to examine whether there is a significant improvement in GAS scores at the end of the year and whether there is a change in students' postsecondary outcomes from end of high school to 3 months out from high school. For the RCT, the research team will use a multilevel model on GAS scores at the end of year and postsecondary outcomes at both post-school time points. Pearson correlations will be used to examine associations in student outcomes and intervention fidelity measures with the CAST participants. Social network analysis will be used to understand integration of services.

Cost Analysis: For the cost analysis, individual ingredients associated with CAST will be identified through a discussion with participants, administrators, and other stakeholders. The costs of each ingredient will then be determined through a review of official records, where possible. Using these various sources, the total cost of implementation will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Students with verified autism and IEPs that designate services for autism
* Caregivers of students with autism
* Special education teachers of students with autism
* Pre-employment specialists of students with autism

Exclusion Criteria:

* Not planning to move or leave their job over the school year

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment of IEP progress (Ruble et al., 2012; 2018). | Outcomes are assessed at the end of the school year (9 months from start of intervention)
  Goal attainment is assessed using psychometric equivalence goal attainment scaling (PET-GAS). Each goal attainment scale used a five-point rating scale: - 2 = student's present levels of performance, - 1 = progress, 0 = expected level of outcome by the end of the school year, +1 = somewhat more than expected, +2 = much more than expected. Half-scores were allowed when raters observed skill levels between two benchmarks. A score of zero represented improvement consistent with the actual description of the written IEP objective. PET-GAS pre- and post-treatment ratings are based on video demonstrations, work samples, and/or data collected by the teacher, caregiver, and/or job coach. In a prior study, two coders independently coded 65% of the goals at baseline and three coders independently rated 35% at final evaluation. Interrater agreement was .94 at baseline and .86 at final evaluation.
Attainment of Postsecondary Goals (Ruble et al., 2019) | Once a year (3 months following school graduation)
  Postsecondary outcomes will be assessed by parent report of attainment in goals (such as enrolling in a training or college program and living independently; Ruble et al., 2019). IEP goal progress is based on a Likert-type scale questionnaire. Parents are asked to think of where the student was at the beginning of the school year with the specific skill (goal) and rate how much progress has been made to date using a five-point scale (1 'none at all' to 5 'a great deal') for each of the three monitored IEP goals. Because CAST prioritizes the development of goals that represent the pivotal areas of instruction for students with autism-social, communication, and learning/work behavior skills, similar goal domains are selected for the control group students for end of the year progress. In a prior study (Ruble et al., 2019), informants' judgments of goal progress were internally consistent across the three goals (alpha) for the parent measure (α = .81) and the teacher measure (α = .69).

SECONDARY OUTCOMES:
Fidelity Assessment of Initial CAST consultation (Ruble et al., 2018) | One time after the initial consultation (within 2 months of the start of the school year).
  Consultant adherence to the initial consultation protocol of CAST is anticipated to be assessed using a 35-item close-ended (yes/no) checklist completed by parents (KR20 = .95), teachers (KR20 = .85), and an independent rater (researcher) (KR20 = .74) (Ruble et al.,2018).
Fidelity Assessment of CAST Coaching (Ruble et al., 2018) | At each coaching session (four timepoints) from fall through spring of school year (about every 4-6 weeks following the initial consulation)
  The second fidelity measure assesses consultant adherence to the coaching protocol. We anticipate using a 17-item checklist (yes/no) completed by teachers and independent raters (KR20 = 1.0) unaware of intervention goals.
Organizational Connectedness | At 2 time points; start of the intervention and at the end of the intervention (over a 9 month period or school year)
  Social network analysis will be used to assess organizational connectedness of team members. Each participant will be asked to identify stakeholders with whom they meet, communicate, actively plan, share information, and collaborate. The purpose is to gather data on directed relational ties between home, school, and community actors involved in the transition process. The relational data will be used to construct and analyze patterns of interaction and service delivery in collaborative networks. For instance, if a school administrator (i) reports trust with a parent (j), but the parent does not report trust with the school administrator, that would indicate the absence of mutual trust. This will also be apparent in the structure of the collaborative network, such as when a directed tie exists from i to j but not from j to i.
Transition Plan Quality (Ruble et al., 2019) | Once per year; at the end of the school year
  Transition Planning Quality (TPQ) will be assessed by parent, teacher, student, and Pre-ETS report. The TPQ is a 30-item four-point Likert parent report scale (1 'strongly disagree' to 4 'strongly agree') that is sensitive to IEP quality and postsecondary outcomes.(Ruble, McGrew, Wong, et al., 2019) The TPQ captures the quality of the transition planning process based on best-practices for transitioning youth, Indicator 13, and focus group results collected from more than 40 stakeholders.(Snell-Rood et al., 2020) Example items are "Students post-high school goals are based on his/her interests and strengths; Student is involved in the decision-making process for his/her education." The internal consistency is .98.(Ruble et al., 2019)

CONTACTS AND LOCATIONS:
Locations (1):
- Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website that explains study and offers assessment tools to use for CAST/COMPASS — http://compassforautism.org